CLINICAL TRIAL: NCT04735588
Title: IMMUNE THROMBOCYTOPENIA (ITP) AND COVID-19: National Retrospective and Prospective Observational Investigation on the Incidence and Course of COVID-19 in Patients With Prior, Ongoing or de Novo ITP. Evaluation of the Impact of COVID-19 Pandemic on the Management of ITP
Brief Title: Investigation on the Incidence and Course of COVID-19 in Patients With Prior, Ongoing or de Novo ITP. Evaluation of the Impact of COVID-19 Pandemic on the Management of ITP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: ITP1021
Record Dates: First submitted 2021-02-02; First posted 2021-02-03 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Immune Thrombocytopenia; ITP; Covid19; ITP Secondary to Infection
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter retrospective and prospective observational study based on the collection of sequential anonymized data from principal Italian ITP centers, to describe the clinical course of ITP patients becoming infected by SARS-CoV-2 and of COVID-19 patients developing de novo ITP.

DETAILED DESCRIPTION:
Multicenter retrospective and prospective observational study based on the collection - through pre-piloted electronic CRFs - of sequential anonymized data from principal Italian ITP centers representative of national geographical distribution, to evaluate, during a 2-years study period, both the cumulative incidence COVID-19 occurring in patients with prior or ongoing ITP (COVID-19 in ITP) and the cumulative incidence of de novo ITP manifesting during COVID-19 (ITP in COVID-19). Data will be collected to describe the clinical course of patients in the two groups. The enrolment period will last 24 months or terminate at the last day of 1-month-COVID-19 free in Italy, whichever comes first. Each patient will be followed up to the first visit scheduled as per common center practice, including at least six months after hospital discharge or end of quarantine home confinement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosed of ITP (ITP could be past, ongoing, persistent >3 months, chronic >12 months) in patients that are in regular follow-up (at least once a year) and who have been diagnosed with COVID-19
* All patients who develop de novo ITP from 1st January 2020 to the end of study after a diagnosis of COVID-19 or during the first 6 months after COVID-19 recovery
* Signed informed consent

Exclusion Criteria:

• All subjects not fitting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ITP becoming infected by SARS-CoV-2 and adult patients with COVID-19 developing de novo ITP, during a study period of two years, starting from 1st January 2020
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Number of ITP patients in which COVID-19 occurs | 24 months
  Cumulative incidence of COVID-19 in adult patients with already known/ongoing ITP
Number of COVID-19 patients developing ITP | 24 months
  Cumulative incidence of adult patients with COVID-19 developing de novo ITP

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - ASST Degli Spedali Civili Di Brescia - UO Ematologia, Brescia
  - Unità di Onco-Ematologia - Azienda Ospedaliera Garibaldi, Catania
  - A.O.U. Careggi - Ematologia, Florence
  - AOU San Luigi Gonzaga - SCDU Ematologia Generale E Oncoematologia, Orbassano
  - Policlinico Universitario Agostino Gemelli, Roma
  - Ematologia Città della Salute e della Scienza di Torino - Molinette, Torino
  - ASST Dei Sette Laghi - UOC Ematologia, Varese
  - AOU Integrata Di Verona, Policlinico G.B. Rossi - UOC Ematologia, Verona